CLINICAL TRIAL: NCT02378675
Title: Influence of the Adipocytokines Apelin, Omentin, Resistin and Visfatin on Lipid Metabolism and Gestational Diabetes Mellitus
Brief Title: Adipocytokines, Gestational Diabetes Mellitus and Lipid Metabolism
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Katharina Worda, Priv. Doz. Dr. Katharina Worda, Medical University of Vienna
Other Study IDs: 11072
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Adipocytokines
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy (1): Adipocytokine levels of patients suffering from GDM are compared to healthy pregnant women
  Interventions: Other: Blood draw
- GDM (2): Adipocytokine levels of patients suffering from GDM are compared to healthy pregnant women
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — During the routine blood sampling, a 10ml plasma sample as well as a 10ml serum sample will be obtained, spinned and stored at -80°C until the final assessment of adipocytokines.

SUMMARY:
Apelin, Visfatin, Omentin and Resistin are adipocytokines derived from human adipose tissue as well as placental tissue and have been shown to be potential mediators of insulin resistance. In each pregnancy, a physiological Insulin resistance syndrome occurs to ensure that the fetus is sufficiently supplied with glucose. Due to their impact on glucose transport mechanisms adipocytokines play an important role for the development of insulin resistance.

Gestational diabetes mellitus (GDM) is one of the most common pregnancy - associated diseases with a prevalence of 5-10% of all pregnancies and its prevalence is increasing. It is associated with severe hazards to both mother and fetus such as macrosomia, plexus palsy, premature delivery and intrauterine death. Furthermore, up to 50% of women with GDM develop Type 2 Diabetes Mellitus (DM2) within the following ten years after pregnancy. GDM seems to be a potent risk factor for the development of DM2 in later life by sharing a number of epidemiological, physiological and genetic characteristics with DM2. Therefore, alterations in adipocytokine levels in women with GDM, if present, may resemble those observed with DM2.

Furthermore, the exact pathogenesis of GDM is not completely understood, however, increased insulin resistance is a well demonstrated mechanism.

Adipocytokines are known to alter insulin resistance through several mechanisms described in the literature. The investigators therefore expect a possible relationship between the above described adipocytokines and gestational diabetes mellitus.

Results of the HAPO-Study have shown a significant association between fetal outcome and mean blood glucose levels in women suffering from GDM. The HAPO Study group supposed a possible relationship between GDM and fetal insulin levels and used C-Peptide to quantify fetal hyperinsulinemia.

A recent study suggests that not only hyperglycemia but also altered maternal lipid metabolism may constitute a risk factor for macrosomia in GDM.

In summary, the investigators aim to illuminate a possible association between the adipocytokines Apelin, Omentin, Resistin and Visfatin, lipid metabolism and gestational diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Informed consent
* Diagnosed gestational diabetes mellitus

Exclusion Criteria:

* Preexisting diabetes mellitus
* Any kind of immunodeficiency
* HIV, HCV, HBV
* Immunomodulating drugs (IF-Gamma, etc.)
* Cancer, chronic diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 150 pregnant women with diagnosed gestational diabetes mellitus (Study group) and 150 pregnant women with normal oral glucose tolerance test (OGTT).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Difference of adipocytokines between women with GDM and women with normal glucose tolerance. | 02/2015

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Worda, Priv.Doz., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria